CLINICAL TRIAL: NCT04479462
Title: The Establishment of Total Joint Arthroplasty Registry Database
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 202001045B0
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Arthritis Knee; Arthritis Hip
MeSH Terms: interventions — Arthroplasty, Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: total joint arthroplasty — The surgery includes primary, revision or partial joint arthroplasty.

SUMMARY:
The purpose of this study will establish total joint arthroplasty registry database in Kaohsiung Chang Gung Memorial Hospital and collect patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary hip or knee arthroplasty
* Patients undergoing revision hip or knee arthroplasty
* Patients undergoing partial hip or knee arthroplasty

Exclusion Criteria:

* Incomplete patients' data
* Follow up less than 1 year after surgery
* Unwillingness to sign the informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include the participants who will receive total joint arthroplasty in our institutte.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Global--10 Score | From the pre-operative assessment until 3 years after the srugery
  Enrolled subjects with total joint arthroplasty of hip and knee will be asked to complete an on-line (web-based) survey (PROMIS-10 global) using a computer. Most patients will only be asked to complete this survey over a maximum 3 year period. The PROMIS-10 Global consists of ten items that measure global physical health (GPH) and general mental health (GMH). The raw PROMIS scores are continuous and range from 4-20. The GPH and GMH scores are converted based on a T-Score Metric allowing for comparisons to a general population. A higher score indicates a better general health
Hip disability and Osteoarthritis Outcome Score, Joint Replacement (HOOS, JR) | From the pre-operative assessment until 3 years after the srugery
  The HOOS, JR is a 6-item instrument that includes 2 of the 5 subscales from the original HOOS (pain, and function and daily living). In the HOOS, JR questionnaire, pain is assessed by 2 items; and function and daily living is assessed by 4 items. These items were assigned a score 0-4 based on the options to the questions (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme). A raw score is summed from the 6 items with a minimum score of 0 and a maximum score of 24. High subscale and raw scores represent worse signs and symptoms. Subsequently, the raw summed score is converted to an interval score out of 100, where 0 represents total hip disability and 100 represents perfect hip health. Using the process, a HOOS, JR score was calculated for each patient included in our study from the original HOOS survey.
Knee injury and Osteoarthritis Outcome Score, Joint Replacement (KOOS, JR) | From the pre-operative assessment until 3 years after the srugery
  The KOOS, JR is a 7-item instrument that includes 3 of the 5 subscales from the original KOOS (symptoms, pain, and function and daily living). In the KOOS, JR questionnaire, stiffness/ symptom is assessed by 1 item; pain is assessed by 4 items; and function and daily living is assessed by 2 items. These items were assigned a score 0-4 based on the options to the questions (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme). A raw score is summed from the 7 items with a minimum score of 0 and a maximum score of 28. High subscale and raw scores represent worse signs and symptoms. Subsequently, the raw summed score is converted to an interval score out of 100, where 0 represents total knee disability and 100 represents perfect knee health. Using the process, a KOOS, JR score was calculated for each patient included in our study from the original KOOS survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No